CLINICAL TRIAL: NCT05429567
Title: Effectiveness of Patient-Controlled Intravenous Analgesia (PCIA) With Fentanyl Background Infusion for Total Hip Replacement
Brief Title: Effectiveness of Patient-Controlled Intravenous Analgesia (PCIA) With Fentanyl
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Collaborators: October 6 University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIRVANA
Record Dates: First submitted 2022-06-19; First posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Total Hip Replacement
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fentanyl infusion Group (Experimental): According to the body weight, 2 ug/kg fentanyl was diluted to 100 ml with normal saline. with rate of 2 mL/h infusions, 10 min lockout time and Initial PCIA analgesia regimen consisting of a 0.5 mL bolus was commenced to be given to the patients postoperative with evaluation the pain
  Interventions: Drug: Fentanyl
- NO fentanyl infusion Group (Experimental): All patients underwent combined spinal and epidural anesthesia (CSEA) with 2 ml of 0.5 % hyperbaric bupivacaine only
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — All patients underwent combined spinal and epidural anesthesia (CSEA) with 2 ml of 0.5 % hyperbaric bupivacaine and 25 ug fentanyl administered using a 27-gauge Whitacre spinal needle and an 18-gauge Tuohy needle in the epidural space. The epidural space was identified utilizing the loss of resistance approach
  Other Names: hyperbaric bupivacaine

SUMMARY:
To enhance post-operative pain management, patient-controlled intravenous analgesia (PCIA) has been employed. The fentanyl background PCIA therapy was created to solve the limitations of IV-based PCIA, such as programming errors, mobility limitations, and the risk of needle stick injuries. The goal of this trial was to observe how fentanyl patient-controlled intravenous analgesia pump (PCIA) and background infusion is worked in patients with post-total hip replacement analgesia.

DETAILED DESCRIPTION:
Significant efforts to enhance the treatment of postoperative pain have resulted in the formulation and implementation of pain management guidelines, as well as the introduction of acute pain services in several hospitals during the last two decades.

Recent research, however, suggests that postoperative pain is still poorly controlled .

Hip replacement procedures are prevalent among the elderly, and they are significantly more painful .

The patient may suffer greatly as a result of the pain, which can also affect physiological functioning caused by hormonal changes caused by sympathetic nervous system activation .

Anaesthesiologists and patients alike are concerned about pain management following major surgery. It should also be mentioned that every pain management medication has certain side effects, especially when an opioid is utilized .

In the clinical ICU, patient-controlled intravenous analgesia (PCIA) has been used to improve postoperative pain management. Titrate analgesics according to demand. It typically provides better pain management and increases patient satisfaction when compared to "on-demand" opioid injections .

The settings programmed into the PCIA machine, such as the bolus dosage, lockout interval, dose restrictions, and background infusion, are included in the PCIA prescription. Each of these factors might have an impact on the safety and efficacy of PCIA.

A new fentanyl-based PCIA therapy has been developed to overcome constraints associated with PCIA provided by IV, such as programming mistakes, mobility limits, and the danger of needle stick injuries.

Prommer and colleagues demonstrated that a fentanyl dosage delivered through PCIA resulted in a mean C max of 1.954 ug/L and a mean absorption of 39.5 ug fentanyl per 10-minute dose delivery time .

ELIGIBILITY:
Inclusion Criteria:

- Patients with total fracture of Hip bones

Exclusion Criteria:

1. History of mental or neurological complaints,
2. Opioid and local anaesthetic allergies,
3. Opioid tolerance,
4. Smoking history,
5. local infection,
6. cemented total hip arthroplasty (THA), revision THA,
7. preoperative DVT,
8. renal failure,
9. bleeding tendency due to anticoagulant therapy

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Fentanyl Background | from 0 hours to 36 hours after the completion of the operation
  Effectiveness of Patient-Controlled Intravenous Analgesia (PCIA) With Fentanyl Background Infusion for Total Hip Replacement

CONTACTS AND LOCATIONS:
Overall Officials: Nirvana Elshalakany, Professor, Principal Investigator — Department of Anesthesia and I.C.U. faculty of Medicine October six university, Egypt
Locations (1):
- October 6 University, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided